CLINICAL TRIAL: NCT01444040
Title: A Prospective, Randomized Evaluation of Subjects With Open-angle Glaucoma, Pseudoexfoliative Glaucoma, or Ocular Hypertension Naïve to Medical and Surgical Therapy, Treated With Two Trabecular Micro-bypass Stents (iStent Inject) or Travoprost Ophthalmic Solution 0.004%
Brief Title: Subjects With Open-angle Glaucoma, Pseudoexfoliative Glaucoma, or Ocular Hypertension Naïve to Medical and Surgical Therapy, Treated With Two Trabecular Micro-bypass Stents (iStent Inject) or Travoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCF-027
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Open-angle Glaucoma
Keywords: Open angle glaucoma; POAG; Ocular hypertension; Pseudoexfoliative glaucoma; Naïve to treatment
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iStent inject (Active Comparator): Implantation of two iStent inject devices
  Interventions: Device: iStent inject
- Drug (Active Comparator): Travoprost drops
  Interventions: Drug: Travoprost

INTERVENTIONS:
Device: iStent inject — Implantation of two iStent inject devices
  Arms: iStent inject
Drug: Travoprost — Travoprost drops
  Arms: Drug

SUMMARY:
Evaluation of the intraocular pressure (IOP) lowering effect of two iStent inject devices versus medical therapy in eyes of subjects with primary open-angle glaucoma, pseudoexfoliative glaucoma, or ocular hypertension naïve to medical and surgical therapy.

DETAILED DESCRIPTION:
Evaluation of the intraocular pressure (IOP) lowering effect of two iStent inject devices versus medical therapy in eyes of subjects with primary open-angle glaucoma, pseudoexfoliative glaucoma, or ocular hypertension naïve to medical and surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Phakic study eye
* IOP ≥ 21 mmHg and ≤ 40 mmHg at the screening visit (subjects with OHT require a second screening IOP measurement

Exclusion Criteria:

* Aphakic or pseudophakic eyes (AC-IOLs or PC-IOLs)
* Previous usage of topical prostaglandin analogues or prior medical therapy for glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Change from screening in mean diurnal IOP (mm Hg) at the Month 12 visit. | 12 months

SECONDARY OUTCOMES:
Change in mean diurnal IOP vs. screening | Month 24
Change in screening in time-wise IOPs | Various Month 12-60
Proportion of responders | Various 12-60 months
  A responder is defined as a subject with a certain target IOP value or a certain reduction of IOP as compared to screening. In the iStent inject group, a responder must not be on an ocular hypotensive medications or have had a postoperative procedure to reposition or remove stent(s) prior to the visit. Due to the lack of a complete consensus on the definition of a clinical responder, a set of target IOP values (e.g., downwards from 22 mm Hg in steps of 1 mm Hg) and reductions of IOP (e.g., downwards from the highest reduction in IOP in steps of 5%) will be evaluated.

OTHER OUTCOMES:
Adverse event reporting | 0-60 months
  Rate of ocular adverse events through 60 months
  * Findings from IOP, best corrected visual acuity, visual field
  * Findings from slit-lamp, fundus and gonioscopic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Lilit A Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Ophthalmological Center, Yerevan, Armenia
Locations (1):
- S.V. Malayan Ophthalmological Center, Yerevan, Armenia